CLINICAL TRIAL: NCT06346171
Title: Evaluating a Virtual Reality Augmented Clinician-Delivered Integrative Psychotherapy Model for Non-Sedated Colonoscopy Procedural Anxiety and Pain: A Prevalidation Trial Protocol (VRIPanx-COL)
Brief Title: VR Augmented Human Delivered Integrative Psychotherapy for Colonoscopy Procedural Anxiety and Pain
Acronym: VRIPanx-COL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Marcel-Alexandru Gaina, MD assist prof Marcel-Alexandru Gaina, Grigore T. Popa University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 408/06.03.2024
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-05

CONDITIONS: Procedural Anxiety; Procedural Pain
Keywords: colonoscopy; anxiety; pain; virtual reality; psychotherapy
MeSH Terms: conditions — Pain, Procedural; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: The VRIPanx-COL study is an RCT investigating the efficacy of VR-facilitated integrative psychotherapy compared to VR distraction only and NSE-Col. Variance minimisation and propensity score matching are used to ensure that the groups are balanced and to supplement the internal validity of evaluating the efficacy of the intervention.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: To ensure credible outcomes, robust blinding for participants, care providers, and outcome assessors is vital to minimize bias. Participants will be briefed generally about participating in VR distraction research, with no details on psychotherapy inclusion. Gastroenterologists and outcome assessors remain blinded to intervention types, using standard tools for unbiased outcome evaluation. The principal investigator, aware of the intervention nature, conducts psychotherapy sessions or engages in simple discussion for control arm VR exposure. Another gastroenterologist oversees randomization to maintain blinding. Standardized VR distractions and pre-programmed randomization ensure unbiased participant allocation, reinforcing study validity through meticulous concealment and blinding protocols.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Virtual Reality Integrative Psychotherapy (Experimental): This group will undergo the same virtual reality exposure software during the colonoscopy procedure, but the psychotherapist will implement the integrative psychotherapy framework during the procedure.
  Interventions: Behavioral: Virtual Reality Integrative Psychotherapy; Device: Virtual Reality Distraction
- Virtual Reality Distraction (Sham Comparator): This group will be exposed to the virtual reality environment as a distraction, but although receiving support in exploring the virtual world, no psychotherapy techniques will implemented.
  Interventions: Device: Virtual Reality Distraction
- Control group (No Intervention): This group will undergo treatment as usual according to state-of-the-art guidelines for non-sedated colonoscopy.

INTERVENTIONS:
Behavioral: Virtual Reality Integrative Psychotherapy — Music therapy: "Weightless" by Marconi Union plays continuously, bridging VR distraction and psychotherapy.
  Before: Patients pick a VR scene (-13 to -10 min), learn VR navigation, and practice 4-7-8 breathing with a VR flower for grounding and resilience (-10 to -9 min). They continue 4-7-8 doing Progressive Muscle Relaxation (4+7 contraction, 8 relaxation), moving from lower body to facial muscles (-8 to -5 min). Values and commitment to action are discussed (-4 to -2 min), emphasizing present-focused thoughts and acceptance (-1 min).
  During: Mindfulness and relaxation are encouraged, with PMR during intense moments. Empowerment and procedural feedback are provided (0 to 30/45 min).
  After: Debriefing normalizes the experience, reinforcing proactive health actions (35 to 50 min).
  Other Names: VRIP
  Arms: Virtual Reality Integrative Psychotherapy
Device: Virtual Reality Distraction — Software: Nature Treks VR nature environments. Hardware: dedicated head-mounted VR display (Oculus Rift S.) powered by a high-end computer (Laptop with at least GTX 1080 graphics card, both with processing units that lower the bottleneck chances); minimum specifications should facilitate presence while limiting cybersickness by ensuring refresh rates beyound 85 frames/second.
  Music therapy: "Weightless" by Marconi Union plays continuously, facilitating sensorial distraction while also allowing blinding.
  Although the psychotherapist will interact with the patient, the dialogue will exclude psychotherapic approaches. The dialogue is designed to be neutral, resembling a comprehensive tutorial for the VR experience. This serves as a comparator to assess the added value of integrating psychotherapeutic techniques within the VR experience.
  Other Names: VRD
  Arms: Virtual Reality Distraction; Virtual Reality Integrative Psychotherapy

SUMMARY:
Colonoscopy is an invaluable tool for the diagnosis and management of colon diseases, especially colorectal cancer (CRC) - the third most common cancer worldwide. Its unmatched ability to detect CRC and premalignant growths makes it the gold standard; however, it is not without its challenges. Patients often experience pre-procedure anxiety and discomfort primarily related to anticipated pain, which negatively impacts both the procedure and its outcomes.

Colonoscopy procedural anxiety not only exacerbates the experience of pain, but also may compromise the quality of bowel preparation, augment procedure and recovery room times, and increase the use of sedation, particularly among females, who report greater pre-procedural anxiety, and perceive the procedure to be more painful and harder to endure. This underscores the importance of interventions aimed at mitigating anxiety to improve patient experience and adherence to colonoscopy procedures.

The profound positive corelation between anxiety and pain impact on outcomes of colonoscopy warrants an investigation of comprehensive patient care strategies. A growing body of evidence indicates that non-pharmacologic interventions, such as music therapy and immersive virtual reality (iVR), may effectively reduce anxiety, pain, and enhance overall patient satisfaction.

Understanding barriers to colonoscopy compliance, such as fear of cancer diagnosis, the perception of invasiveness, and feelings of embarrassment is paramount to enhancing CRC screening uptake, therefore lowering mortality.

DETAILED DESCRIPTION:
The proposed VR-Facilitated Integrative Psychotherapy framework (VRIPainX-COL) leverages the immersive capabilities of VR as platform fir psychological interventions for this pilot trial is designed to assess its preliminary efficacy, acceptability, and feasibility in reducing the pre-procedural anxiety and discomfort associated with colonoscopy.

Primary Aims:

1.1 Developing a comprehensive conceptual framework for colonoscopy procedural anxiety and pain reduction through a a humanised digital interface using virtual reality distraction as platform for integrative psychotherapy support VRIPanx-COL; 1.2 Clinically implementing the VRIPanx-COL blueprint within a methodological design aimed at assessing its preliminary efficacy in reducing perceived procedural anxiety and pain compared to 1.3 VR distraction alone and 1.4 conventional non-sedated colonoscopy

Secondary Aims:

2.1 Evaluate the feasibility and acceptability of implementing VRIP-Col interventions during non-sedated colonoscopy, 2.2 Gathering qualitative feedback from both patients and performing colonoscopists regarding VRIP experienced advantages, obstacles and their perspectives for enhancing the intervention.

ELIGIBILITY:
Inclusion criteria:

* scheduled non-sedated colonoscopy.
* cognitive ability to understand study aims;
* willingness to participate and provide written consent.

Exclusion criteria:

* emergency colonoscopy;
* significant sensory-cognitive impairments;
* potential risk of:

  1. photic seizures;
  2. photosensitivity;
  3. severe motion sickness;
  4. allergies to materials used.
* anxiety disorders:

  1. use of psychoactive or analgesic substances;
  2. concomitant psychotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Available to individuals of all self-identified genders, with endeavours to equilibrate representation across cohorts to acquire comparative insights concerning the reported vulnerability of the biological female sex to anxiety, pain, and discomfort.
Enrollment: 36 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Procedure-Related Anxiety | STAY-Y1: baseline anxiety measured within 20 minutes before the procedure; post-procedural anxiety (within 20 minutes after the procedure's completion).
  This measure assesses the degree of reduction in anxiety related to undergoing a non-sedated colonoscopy procedure. Anxiety levels will be quantified using the Spielberger STAI-Y1 and STAI-Y2 forms, previously standardized to the Romanian population and approved by Romanian Psychological College. STAI-Y1 and Y2 are applied and interpreted by a licensed investigator, in order to ensure viability of collected data. The scale measures how respondents feel at a particular moment in time and in general, providing insight into both state and trait anxiety levels. The difference in STAI-Y1 scores from baseline (pre-intervention) to post-procedure will be analyzed to determine the effectiveness of the VR-Augmented Integrative Psychotherapy in reducing procedural anxiety compared to Sham VR Distraction and control groups.
Pain perception | Within 20 minutes before the colonoscopy procedure (baseline) and immediately after the procedure (within 20 minutes post-procedure).
  The primary measure of pain perception will be the Visual Analog Scale (VAS), a validated tool for pain assessment. This self-reported measure allows patients to rate their pain on a scale from "no pain" (0) to "worst imaginable pain" (10).

SECONDARY OUTCOMES:
Feasibility and Acceptability of VRIP-Col Interventions | Data on feasibility and acceptability will be collected within 24 hours after the colonoscopy procedure.
  This outcome will assess the logistical feasibility and overall acceptability of the VRIP-Col interventions among patients undergoing non-sedated colonoscopy. Feasibility metrics will include the successful integration of VRIP-Col into clinical workflows, the ability to deliver the intervention to all enrolled participants without disrupting standard care procedures, and the technical reliability of VR equipment. Acceptability will be evaluated through patient and healthcare provider satisfaction surveys, focusing on the perceived usefulness, ease of use, and willingness to use or recommend the VRIP-Col interventions in the future.
Qualitative Feedback on VRIP-Col Interventions | Data on feasibility and acceptability will be collected within 24 hours after the colonoscopy procedure.
  This outcome will involve the collection and analysis of qualitative feedback from patients who receive the VRIP-Col interventions and the colonoscopists who perform the procedures. Feedback will be gathered through semi-structured interviews designed to explore the perceived advantages of the VRIP-Col interventions, any obstacles encountered during their implementation, and suggestions for improvement from both the patient and provider perspectives. This qualitative analysis will provide insights into the user experience, identify potential barriers to effective implementation, and inform future refinements of the VRIP-Col approach.

OTHER OUTCOMES:
Trait anxiety | Within 72 hours after study enrolment.
  STAI-Y2 will reveal the participants general anxiety in order for a more relevant group matching. Participants general tendency to perceive and respond to situations as threatening or anxiety-inducing. It will be applied after enrolling.
Quality of Life impact VRIP-Col | Within 36 hours before and after the colonoscopy procedure.
  Assessment of the bio-psycho-social interplay of VRIP as reflected by the score dynamic of the Health, Self-Esteem, relationships and Goals and Values items assessed by a qualified researcher using a Romanian population-standardised Quality of Life Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel A Gaina, ass.prof. MD, Study Director — University of Medicine and Pharmacy "Grigore T Popa" Iasi, Romania; Cristinel Stefanescu, Prof. MD, Study Chair — University of Medicine and Pharmacy "Grigore T Popa" Iasi, Romania
Locations (1):
- University of Medicine and Pharmacy Grigore T Popa, Iași, Iaşi, Romania

IPD SHARING:
Plan to Share IPD: Yes
Following the conclusion and dissemination of the primary results of our study, we are committed to sharing the IPD and its supplementary documentation - including the study protocol, statistical analysis plan, informed consent form, and the clinical study report - with qualified investigators bestowing a scientifically valid analysis proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning at a juncture of six months succeeding the disclosure of the principal results, the datasets will remain accessible for a span of three years. This provisional period is established to facilitate expedited access to data while preserving the sanctity of ongoing analyses and proprietary knowledge.
Access Criteria: This framework is intended, in part, to allow immediate and early data access, while also preserving the privacy of concurrent analyses and integrity of intellectual property. mplementation of successful proposal submission for any qualified investigator with a scientifically valid and beneficial proposal for solving a significant provider or patient health issue based directly on the primary research questions or the study objectives. A specially constituted and independent review panel of external scientific experts and research experts will evaluate the submitted proposals. Data use agreement: A basic agreement declaring the responsible and ethical use of the data and requiring the investigators to certify privacy protocols and to safeguard patient-specific information.

REFERENCES:
- [Background] Gaina MA, Szalontay AS, Stefanescu G, Balan GG, Ghiciuc CM, Bolos A, Gaina AM, Stefanescu C. State-of-the-Art Review on Immersive Virtual Reality Interventions for Colonoscopy-Induced Anxiety and Pain. J Clin Med. 2022 Mar 17;11(6):1670. doi: 10.3390/jcm11061670. PMID 35329993